CLINICAL TRIAL: NCT02614105
Title: UriCO - Effect of Pelvic Floor Muscle Training and Cough-suppression Therapy on Urinary Incontinence Amongst Women With Chronic Obstructive Pulmonary Disease; a Randomised Controlled Trial
Brief Title: Urinary Incontinence Amongst Women With Chronic Obstructive Pulmonary Disease
Acronym: UriCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Stacey Haukeland Parker, MSc/senior physiotherapist, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3342
Record Dates: First submitted 2015-11-16; First posted 2015-11-25 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Urinary Incontinence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pelvic floor muscle training (Experimental): Participants in the pelvic floor muscle training group will receive group exercise sessions (1 hour) at the physiotherapy out-patient department of the hospital once a week for 16 weeks with guidance from an experienced pelvic floor physiotherapist. The group exercise sessions will focus on pelvic floor muscle training, relaxation and breathing techniques. Participants in the pelvic floor muscle training group will also receive an individually adapted pelvic floor muscle training program for daily home use.
  Interventions: Procedure: Pelvic floor muscle training
- Cough-suppression (Experimental): Participants in the cough-suppression group will receive a group education session with general information about cough-suppression therapy and advice about how to distinguish between unproductive and productive cough to enable them to perform airway clearance techniques when required. In addition, participants will receive one to two individual sessions (30-60 minutes) of cough-suppression therapy tailored to the individual needs based on symptoms and underlying disease activity
  Interventions: Procedure: Cough-suppression therapy
- Control group (Experimental): Participants in the group will receive guidance and instruction in terms of correct contraction of the pelvic floor muscles at clinical assessment. Control group participants will receive brief written information about pelvic floor muscle training and cough-suppression therapy, but no other form of regular follow-up or intervention throughout the intervention period.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Pelvic floor muscle training — 16 weeks of group-based exercise
  Arms: Pelvic floor muscle training
Procedure: Cough-suppression therapy — Group and individual sessions of respiratory physiotherapy with focus on techniques to suppress cough
  Arms: Cough-suppression
Other: Control — Brief information only
  Arms: Control group

SUMMARY:
The primary aim of the study is to investigate whether pelvic floor muscle training or cough-suppression therapy reduces symptoms of urinary incontinence amongst women with chronic obstructive pulmonary disease grade 1-4 (mild to very severe disease).

DETAILED DESCRIPTION:
This two-centre study will consist of a randomised controlled trial (RCT) with a parallel group design and include two intervention groups and one control group. Recruitment and data collection will occur simultaneously at the ØHT and St. Olav's Hospital in Trondheim.

All participants will complete an initial four week general group exercise class (1 hour once a week) prior to randomisation. This intervention will focus on strength exercises (lower limb and upper limb), endurance training, balance training and thorax mobilising exercises. All participants will be examined and complete questionnaires at two occasions; after the initial four weeks general exercise/before intervention, and at 16 weeks post-randomisation.

Participants will be randomised to either Intervention group A (pelvic floor muscle training group), Intervention group B (cough-suppression group) or a control group who will receive brief written information about pelvic floor muscle training and cough-suppression, but no other form of regular follow-up or intervention throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* COPD grade 1-4
* Subjective urinary incontinence
* Ability to perform an active contraction of the pelvic floor muscles

Exclusion Criteria:

* Unstable COPD
* More than 4 hospital admissions due to COPD in the past twelve months
* Neurological conditions
* Previous gynecological surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short form (ICIQ_SF) | Change from baseline score at 16 weeks
  Participants in the group will receive guidance and instruction in terms of correct contraction of the pelvic floor muscles at clinical assessment. Control group participants will receive brief written information about pelvic floor muscle training and cough-suppression therapy, but no other form of regular follow-up or intervention throughout the intervention period.

SECONDARY OUTCOMES:
Cough symptoms | Change from baseline score at 16 weeks
  Cough symptoms will be measured using the Norwegian version of the Leicester Cough Questionnaire, which is in the process of being translated from English to Norwegian and tested for reliability and validity. The Leicester Cough Questionnaire is used to measure physical, psychological and social factors related to cough
Chronic Obstructive Pulmonary Disease symptoms | Change from baseline score at 16 weeks
  A subjective evaluation of their Chronic Obstructive Pulmonary Disease symptoms (including cough) using the COPD Assessment Test (CAT). CAT is a disease-specific questionnaire which measures subjective symptoms of Chronic Obstructive Pulmonary Disease.
Self-reported function and quality of life | Change from baseline score at 16 weeks
  COOP/WONCA is quick and easy to complete and has demonstrated good validity and reliability both in Norwegian and in the Chronic Obstructive Pulmonary Disease population
Voluntary pelvic floor muscle function | Change from baseline score at 16 weeks
  Voluntary pelvic floor muscle function will be evaluated using digital palpation and scored on a 1-4 scale according to the International Continence Society Score.
Pelvic floor muscle strength | Change from baseline score at 16 weeks
  Pelvic floor muscle strength will be measured using Peritron.
Field walking test | Change from baseline score at 16 weeks
  Participants will also perform the six-minute walk test at inclusion and after the intervention to explore whether the intervention results in a change in general physical capacity.
Physical activity | Change from baseline score at 16 weeks
  Physical activity will be measured using an activity monitor (pedometer) which the participants will wear throughout the whole intervention period to investigate whether a change in urinary incontinence affects physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Hege Hølmo Johannessen, PhD, Principal Investigator — Ostfold Hospital
Locations (2):
- Norway (2):
  - St Olavs Hospital, Trondheim
  - Østfold Hospital Trust, Moss, Østfold fylke

REFERENCES:
- [Derived] Haukeland-Parker S, Frisk B, Spruit MA, Stafne SN, Johannessen HH. Treatment of urinary incontinence in women with chronic obstructive pulmonary disease-a randomised controlled study. Trials. 2021 Dec 11;22(1):900. doi: 10.1186/s13063-021-05816-2. PMID 34895285